CLINICAL TRIAL: NCT01081392
Title: The Role of Inhaled Particle Size on the Inflammatory Response Induced by Endotoxin Inhalation
Brief Title: Inflammatory Markers in Sputum After LPS Inhalation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Brugmann (Other)
Responsible Party: Jean-Pierre Tassignon, MD, PhD, Head Clinical Research Unit, CHU Brugmann
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CIA-01.2
Record Dates: First submitted 2010-03-02; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Inflammation
Keywords: LPS; endotoxin; inflammatory markers; healthy volunteers; neutrophils in sputum
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- LPS sequence 1 (Experimental): Nebulizers A then B then C
  Interventions: Biological: LPS
- LPS sequence 2 (Experimental): Nebulizers B then C then A
  Interventions: Biological: LPS
- LPS sequence 3 (Experimental): Nebulizers C then A then B
  Interventions: Biological: LPS
- LPS sequence 4 (Experimental): Nebulizers A then C then B
  Interventions: Biological: LPS
- LPS sequence 5 (Experimental): Nebulizers C then B then A
  Interventions: Biological: LPS
- LPS sequence 6 (Experimental): Nebulizers B then A then C
  Interventions: Biological: LPS

INTERVENTIONS:
Biological: LPS — LPS 20mcg sd inhaled via nebulizer, 3 periods

SUMMARY:
The purpose of the study is to measure inflammatory biomarkers in sputum and peripheral blood in healthy volunteers after inhalation of single doses of LPS (20 mcg) administered as particles of different sizes.

DETAILED DESCRIPTION:
Endotoxins are inflammatory substances present in the environment. In man, the inhalation of the lipopolysaccharride moiety (LPS) induces measurable immune responses. With an inhaled single dose of 20 micron, the inflammatory response in man is sub-clinical. During bronchoprovocation tests with allergens, the particle size determines to a large extent the intensity of the response. the response to LPS as a function of particle size is not known and will be studied in this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer, non-smoking or ex-smoker >1mth and <10packs/year
* normal ECG
* normal lab values for hematology, ionogram, AST, ALT, alk phosphatases, urea, creatinine and CRP
* FEV1/forced vital capacity >0.7 and FEV1>80% of predicted value
* able to produce valid sputum following induction (>=50% viable cells, <50% squamous cells and <60% neutrophils)
* females must be using contraception
* written informed consent

Exclusion Criteria:

* infection within 14 days
* history of bronchial asthma
* obstructive respiratory condition with FEV1 <70% of theoretical value

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Absolute neutrophil count in sputum | 24hrs after LPS inhalation

SECONDARY OUTCOMES:
white blood cells and differential in peripheral blood | 0, 6 and 24 hrs after LPS inhalation
CC16 in peripheral blood | 0, 6 and 24hrs after LPS inhalation
Calgranulin A/B | 0, 6 and 24hrs after LPS inhalation
CRP in peripheral blood | 0, 6 and 24hrs after LPS inhalation
Spirometry (FEV1 and FEV1/FEV) | 0, 1, 6 and 24hrs after LPS inhalation
Alveolo-capillary diffusion | 0, 6 and 24hrs after LPS inhalation
12-lead ECG | Screening Visit 1 and final Visit 5
Physical exam | At the Screening Visit 1, at the three Visits with LPS inhalation and at the Final Visit
  A complete physical exam at screening and at the final Visits, and an abbreviated physical exam at the three Visits during which LPS will be administered
Safety labs from peripheral blood | At the Screening Visit 1 and the Final Visit 5
  hematology, blood chemistry (ionogram, AST, ALT, alkaline phosphatases, urea, creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MICHEL, MD, PhD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Derived] Doyen V, Pilcer G, Dinh PH, Corazza F, Bernard A, Bergmann P, Lefevre N, Amighi K, Michel O. Inflammation induced by inhaled lipopolysaccharide depends on particle size in healthy volunteers. Br J Clin Pharmacol. 2016 Nov;82(5):1371-1381. doi: 10.1111/bcp.13052. Epub 2016 Jul 28. PMID 27331367